CLINICAL TRIAL: NCT05003414
Title: A Prospective, Multicentre, International, Post-marketing, Longitudinal, Observational Cohort Study to Monitor the Performances of GMK Sphere Cementless Knee Prosthesis
Brief Title: The Medacta International GMK Sphere Cementless Post-Marketing Surveillance Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P02.014.26
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Arthritis; Traumatic Arthritis; Rheumatoid Arthritis; Poly-arthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: GMK Sphere cementless Knee Replacement — Performance of Total Knee Arthroplasty (TKA) with GMK Sphere cementless Knee Replacement

SUMMARY:
This is a Post-Marketing Surveillance study of GMK Sphere cementless knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* A disabled or severely disabled joint as a result of arthritis, traumatic arthritis, rheumatoid arthritis, poly-arthritis or avascular necrosis
* Patients between the age of 18 and 80 at the time of consent
* Listed for total knee replacement surgery.
* Patients who are willing and able to give informed written consent

Exclusion Criteria:

* Progressive local or systemic infection
* Muscular loss, neuromuscular disease or vascular deficiency of the affected limb, making the operation unjustifiable
* Severe instability secondary to advance destruction of condralar structures or loss of integrity of the medial or lateral ligament
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems
* Patient whose BMI exceeds 40
* Any case not described in the inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring Total Knee Arthroplasty and who are suitable to receive Medacta GMK Sphere cementless Knee Replacement will be proposed to take part to the current post-market surveillance study during their pre-operative visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 10 years
  Kaplan Meier method

SECONDARY OUTCOMES:
Clinical outcome: Knee Society score | Preop and 1, 2, 5, 10 years postop
  Knee Society Score (KSS): evaluates pain, in a total of 50 points, stability, 25 points, and range of motion, 25 points. The maximum score of 100 points is reached when there is no pain, with good alignment of the knee in extension, and at least 125° of range of motion, without any anteroposterior or mediolateral instability.
Patient-reported outcome: Forgotten Joint Score | 1, 2, 5, 10 years postop
  Forgotten Joint Score (FJS) is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment.It consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities
Radiographic performance of the implants looking for radiolucencies, migration, loosening, subsidence | Immediately postop + 1, 2, 5, 10 years postop
  Presence of radiolucencies, migration, loosening, subsidence
Intraoperative and postoperative Adverse events | Intraop + Immediately postop + 1, 2, 5, 10 years postop
  Intraoperative and postoperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Marchetti, MD, Principal Investigator — Clinique Saint Vincent de Paul
Locations (5):
- France (4):
  - Clinique Saint Vincent de Paul, Bourgoin
  - Clinique du Parc, Caen
  - Hôpitaux Civils de Colmar, Colmar
  - Clinique des Acacias, Cucq
- Hôpital de la Tour, Meyrin, Switzerland

IPD SHARING:
Plan to Share IPD: No